CLINICAL TRIAL: NCT02103790
Title: Installation of Non-invasive Ventilation at Home Using Telemedicine : a Pilot Study on Feasibility and Impact on Ventilation Compliance
Acronym: Tele-VAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Principal Investigator, david orlikowski, coordinating physician - professor, Centre d'Investigation Clinique et Technologique 805
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-A01817-38
Record Dates: First submitted 2014-04-01; First posted 2014-04-04 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Neuromuscular Diseases; Kyphoscoliosis; Non Invasive Ventilation
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Home NIV installation (Experimental)
  Interventions: Device: Home NIV installation

INTERVENTIONS:
Device: Home NIV installation

SUMMARY:
Neuromuscular diseases are frequently associated with respiratory failure, which requires Non Invasive Ventilation (NIV). Currently, the NIV installation is done during an hospitalization of several days. This hospitalization is problematic because of availability of beds, logistical difficulties for the patient and estrangement from the usual environment.

For this reasons, the NIV installation at home could be an interesting alternative for both the patient and the medical staff.

The aim of this pilot study is to test the feasibility of NIV installation at home, using telemedicine as a remote monitoring tool, and to assess its impact on the ventilation compliance.

DETAILED DESCRIPTION:
For the study protocol, patients will be hospitalized for the first day to define the ventilation mode and initial parameters, and to choose the best adapted interface.

Then, the patient is discharged from hospital and parameters adaptation is continued at home during the following five days by the hospital medical staff, using telemedicine. An ASV Santé employee visits the patient at home everyday during 5 days to ensure follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Man or Women aged over 18 years
* Neuromuscular disease or kyphoscoliosis
* At least one sign among : dyspnea, orthopnea, daytime sleepiness, cephalalgia, asthenia
* At least one sign among : hypercapnia > 45 mmHg, desaturation time < 88%, night desaturation time > 5 min, Vital Capacity < 60% or Pimax < 60 cm H2O.

Exclusion Criteria:

* Mechanic ventilation refusal
* Patient living alone
* Acute respiratory failure
* Patient who need a third party for the ventilation installation
* Severe respiratory limitation
* Home oxygen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Number of required days to obtain a 4-hours-night ventilation | 5 days

SECONDARY OUTCOMES:
Number of ventilation hours per 24 hours during the 5 first days | 5 days
Capno-oximetry improvement at D5 | 5 days
Capno-oximetry and arterial blood gases improvement at D30 | 30 days
Clinical signs decrease (symptoms, dyspnea, drowsiness) | 30 days
Number of non programmed home visits | 5 days
Economic cost evaluation | 5 days
Number of skin slough caused by interface position | 30 days
Number of hospitalization for respiratory or ventilation disorder | 30 days
Satisfaction scale for the patient and his family at D5 and D30 | 30 days
  CSQ8 and VAS (Visual Analogical Scale)
Quality of life (SF36) at D1 and D30 | 30 days
Reliability of telemonitoring | 5 days
  Cross between ventilation parameters read remotely and ventilation parameters audited at patient home (by an ASV Santé employee)
Reliability of telemedicine | 5 days
  Cross between ventilation parameters modified remotely and ventilation parameters audited at patient home (by an ASV Santé employee)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Raymond Poincaré, Garches, France